CLINICAL TRIAL: NCT01225705
Title: An Open, Prospective Study to Compare the Safety and Efficacy of Raltegravir vs. Atazanavir / Ritonavir, Both in Combination With Tenofovir DF and Emtricitabine, in the Treatment of HIV-infection in ART Naive Subjects With HCV Co-infection.
Brief Title: Safety Study of Raltegravir in HIV/HCV Co-infected Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no pts recruited
Sponsor: University Hospital, Bonn (Other)
Collaborators: Dr. Axel Baumgarten, Berlin (Unknown); Dr. Christoph Stephan, Frankfurt/M (Unknown); Dr. Stefan Esser, Essen (Unknown); Dr. Keikawus Arastéh, Berlin (Unknown); Prof. Dr. Hans-Jürgen Stellbrink, Hamburg (Unknown); Dr. Thomas Lutz, Frankfurt/M (Unknown); Dr. Jörg Gölz , Berlin (Unknown)
Responsible Party: Rheinische Friedrich-Wilhelms-Universität Bonn, Germany, Bonn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKB-2009-MED-I-JKR-01; 2009-015904-24 (EudraCT Number)
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-10

CONDITIONS: HIV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Raltegravir Potassium; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir (Experimental): 45 patients will receive open label raltegravir, in addition to the common backbone tenofovir and emtricitabine
  Interventions: Drug: raltegravir
- Atazanavir/ritonavir (Active Comparator): 45 patients will receive open label atazanavir/ritonavir
  Interventions: Drug: Atazanavir/ritonavir

INTERVENTIONS:
Drug: raltegravir — Patients will be randomized 1:1 to either the experimental or the active control arm
  Arms: Raltegravir
Drug: Atazanavir/ritonavir — Patients will be randomized 1:1 to either the experimental or the active control arm
  Arms: Atazanavir/ritonavir

SUMMARY:
Current European AIDS Clinical Society (EACS) guidelines for the treatment of HIV infection recommend a combination antiretroviral regimen composed of two nucleoside reverse transcriptase inhibitors plus a ritonavir boosted protease inhibitor or a non-nucleoside reverse transcriptase inhibitor.

The non-nucleoside reverse transcriptase inhibitors licensed for naïve patients - nevirapine and efavirenz - have both been asociated with increased rates of hepatotoxicity (nevirapine) and CNS toxicity (efavirenz) in HIV/HCV co-infected patients. Although PI-based therapy has dramatically reduced morbidity and mortality, it has been limited by complex dosing regimens and toxicities, leading to adherence challenges. Varying degree of liver insufficiency may necessitate pharmacokinetic monitoring of the protease inhibitor and may necessitate dose adjustments. In HIV/HCV co-infected patients HAART based on another class of antiretrovirals than NNRTI or PI may thus offer advantages with regard to adverse events and thus long-term efficacy.

The overall intention of this trial is to examine in a non-inferiority design the safety and efficacy of a raltegravir based HAART with a standard-of-care HAART in HIV-/HCV co-infected patients. The standard of care used in this study will be atazanavir/ritonavir. All patients will in addition receive a fixed combination of tenofovir and emtricitabine.

The primary end-point is the rate of hepatotoxic events, defined by ALT elevations.

ELIGIBILITY:
Inclusion Criteria:

* HIV and Hepatitis C co-infected patients
* indication for HAART according to current German-Austrian guidelines
* HAART naive
* no primary NRTI / Integrase / PI associated resistance mutation according to the Stanford algorithm at screening; every patient MUST have a genotypic resistance assay prior baseline available (< 6 months prior to baseline)
* women of childbearing age: negative pregnancy test
* ability to sign written informed consent

Exclusion Criteria:

* advanced liver cirrhosis Child-Pugh B or C or decompensated liver disease
* Pegylated interferon / ribavirin or other anti-HCV therapy; planned anti-HCV therapy for duration of the study (48 weeks).
* acute or chronic hepatitis B infection
* acute hepatitis A or other hepatotropic virus infections
* any other chronic liver disease such as alcohol abuse or hemosiderosis
* use or planned use (for the duration of the study, 48 weeks) of rifampicin, St. John´s wort and drugs that are metabolized via the cytochrome P450 system with a narrow therapeutic PK-range such as astemizole, terfenadine, cisapride, pimozide, chinidin, bepridil, triazolam, midazolam, ergotamine, dihydroergotamin, ergometrine, methyl-ergometrine. FOR OTHER COMEDICATIONS please consult with the SPC of Raltegravir (Isentress®), Atazanavir (Reyataz®), Ritonavir (Norvir®), your hospital pharmacist, www.hiv-drug-interactions.org or the principal investigator in case of uncertainty.
* new AIDS defining event, except for Kaposi sarcoma, < 1 months prior to screening
* malignancy, except for Kaposi sarcoma, with current radio- or chemotherapy
* history of organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Primary objective
  1. there is no difference in the rate of grade 1/2, or 3/4 ALT elevations
  2. there is a higher incidence of grade 1 - 4 hyperbilirubinemias in the ATV/r arm

SECONDARY OUTCOMES:
Secondary objectives
  Other parameters of safety and efficacy will be compared between both arms

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - Auguste Viktoria Hospital (AVK), Berlin
  - Praxiszentrum Kaiserdamm, Berlin
  - Private Practice Dupke, Carganico, Baumgarten, Berlin
  - Department of Internal Medicine I, Bonn University, Bonn
  - University of Essen, Essen
  - Infektiologikum Frankfurt, Frankfurt am Main
  - University of Frankfurt, Frankfurt am Main
  - Infektionsmedizinisches Centrum Hamburg (ICH), Hamburg